CLINICAL TRIAL: NCT06984666
Title: The Perception of Lower Third of the Face Combined With Digital Virtual Models and the Clinical Phenotype at 45° Viewing Angle : a Clinical Study
Brief Title: Facial Aesthetic Analysis Model Based on Clinical Cohort Phenotype to Explore 45° Facial Profile.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Linyu Xu (Other)
Collaborators: Stomatological Hospital Affiliated with Fujian Medical University (Other)
Responsible Party: Sponsor-Investigator, Linyu Xu, Director of the Department of Orthodontics at the Stomatological Hospital Affiliated with Fujian Medical University, Stomatological Hospital Affiliated with Fujian Medical University
Organization: Stomatological Hospital Affiliated with Fujian Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024Clin003
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-09

CONDITIONS: Malocclusion, Angle Class II; Malocclusion, Angle Class III
Keywords: Midface; Eye tracking; Aesthetic evaluation; Perception; morphology
MeSH Terms: conditions — Malocclusion, Angle Class II; Malocclusion, Angle Class III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Free browsing (No Intervention): This phase of the experiment serves as baseline data without language intervention.
- Language cue (Experimental): In this phase of the experiment, participants are given language cues to intervene in their eye movement.
  Interventions: Behavioral: language

INTERVENTIONS:
Behavioral: language — Language cues are used to provide participants with psychological suggestions in order to achieve the goal of shifting their focus in gaze patterns.
  Arms: Language cue

SUMMARY:
Facial aesthetics has always been a complex and subjective concept. The overall facial harmony, along with lip protrusion, which is often a focus for orthodontists, requires evaluation from multiple perspectives. The viewing angle also influences the assessment of facial aesthetics, particularly the judgment of lip protrusion. This study aims to explore the differences in facial fixation patterns and aesthetic evaluations among different populations at specific viewing angles by using digital models to simulate various perspectives.

DETAILED DESCRIPTION:
In the analysis of facial aesthetics, the 45° profile has a unique advantage in evaluating lip protrusion, zygomatic fullness, and contour curve. Compared to the frontal view, this angle provides a more three-dimensional and deeper perspective. In a previous study, the research group found that the shape of the midface area at 45° influences the evaluation of lip protrusion. In this study, a digital model was used to simulate the protrusion of different midface areas in order to explore the differences in facial fixation patterns and aesthetic evaluations among various individuals at 45°. Based on data from individuals who showed significant improvement in frontal and profile beauty before and after clinical treatment, the study added an evaluation of beauty and lip position from the 45° profile. This aims to provide a reference for the subsequent establishment of a 45° profile analysis.

ELIGIBILITY:
Inclusion Criteria:

Orthodontist inclusion criteria: ① With dental doctor qualification certificate; ② At least 2 years of professional training in orthodontics.

Inclusion criteria for orthodontic patients: ① Receiving orthodontic treatment for more than 1 year; ② Volunteer to participate in the study; ③ Native language is Chinese, can understand the prompt language and normal communication.

General adult inclusion criteria: ① have not experienced orthodontic treatment or have no need for orthodontic treatment; ② Do not engage in stomatology industry, have not studied stomatology specialty; ③ Native language is Chinese, can understand the prompt language and normal communication.

Exclusion Criteria:

① have visual impairment (such as color blindness, high myopia); ②Have psychological problems (such as autism, schizophrenia); ③ Recent use of alcohol, or long-term fatigue, anxiety; Current use of any medication that may affect cognitive ability; ⑤ Use mascara, contact lenses or small frame height glasses

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Total fixation duration of area of interest | The duration of the experiment for each participant does not exceed 10 minutes. A random selection of 10 participants will immediately undergo a repeat experiment after the first round to verify the reliability of the participants.
  The facial images used as stimulus materials are divided into several regions, with the fixation duration in each area of interest serving as the primary measurement. Changes in fixation duration represent a shift in the focus of attention.

SECONDARY OUTCOMES:
Eye movement track | The duration of the experiment for each participant does not exceed 10 minutes.A random selection of 10 participants will immediately undergo a repeat experiment after the first round to verify the reliability of the participants.
  The specific patterns of attention shift will be further observed through the changes in eye-tracking trajectories.

CONTACTS AND LOCATIONS:
Locations (1):
- Stomatological Hospital Affiliated with Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
There are concerns about excessive patient privacy intrusion, and some patients are unwilling to provide all the requested information, such as unmasked facial data and other sensitive details.